CLINICAL TRIAL: NCT00254072
Title: Evaluation of Endostapled Anastomoses for Laparoscopic Gastric Bypass (EEA-LGB)a Prospective Randomized Comparison of the 3.5 mm vs 4.8 mm Circular Stapler for Creation of the Gastrojejunostomy in Prevention of Staple Line Hemorrhage During Laparoscopic Gastric Bypass
Brief Title: Evaluation of Endostapled Anastomoses for Laparoscopic Gastric Bypass (EEA-LGB)
Acronym: EEA-LGB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: United States Surgical Corporation (Other)
Responsible Party: Ninh T. Nguyen, MD /Chief, Division of Gastrointestinal Surgery, University of California, Irvine Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS 2005 4474; SPA 38461
Record Dates: First submitted 2005-10-31; First posted 2005-11-15 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Morbid Obesity
Keywords: Morbid Obesity; Laparoscopic Gastric Bypass; Staple Line Hemorrhage
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smaller Stapler (Active Comparator): 3.5 mm Circular Stapler
  Interventions: Procedure: 3.5 mm vs 4.8 mm Stapler During Laparoscopic Gastric Bypass
- Larger Stapler (Active Comparator): 4.8 mm Circular Stapler
  Interventions: Procedure: 3.5 mm vs 4.8 mm Stapler During Laparoscopic Gastric Bypass

INTERVENTIONS:
Procedure: 3.5 mm vs 4.8 mm Stapler During Laparoscopic Gastric Bypass — The procedure consists of a creation of a small gastric pouch and rerouting the small bowel to bypass the stomach and duodenum. There are two anastomoses in this procedure: the gastrojejunostomy and the jejunojejunostomy.
  Other Names: Covidien small 3.5 mm Circular Stapler; Covidien large 4.8 mm Circular Stapler

SUMMARY:
Laparoscopic gastric bypass surgery is a common procedure being performed for the treatment of morbid obesity. The procedure consists of a creation of a small gastric pouch and rerouting the small bowel to bypass the stomach and duodenum. There are two anastomoses in this procedure: the gastrojejunostomy and the jejunojejunostomy. Potential complications after gastric bypass include gastrointestinal bleeding and leaks. Gastrointestinal bleeding can occur at any staple line including the gastrojejunostomy. Potential methods for prevention of postoperative gastrointestinal bleeding include oversewing of the anastomosis or the use of a smaller stapler height. We hypothesize that the use of staplers with smaller staple height will significantly result in a lower rate of staple line bleeding and possible leaks.

DETAILED DESCRIPTION:
RATIONALE:

1. Gastrointestinal (GI) bleeding can occur in up to 4% of cases. GI bleeding is associated with significant morbidity which may include transfusion and possible re-operation
2. Leaks at the gastrojejunostomy can be potentially life threatening and ranged from 1% to 2%.

HYPOTHESES:

The smaller circular stapler may be associated with a lower rate of intraoperative intraluminal bleeding and postoperative gastrointestinal bleeding than the larger one.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 40-60 kg/m2
2. BMI of 35 kg/m2 with comorbidities

Exclusion Criteria:

1. large abdominal ventral hernia
2. large hiatal hernia,
3. history of liver cirrhosis
4. history of venous thrombosis or pulmonary embolism, coagulopathy or
5. Pregnant women

   * All physician, hospital, surgery, and laboratory costs will be billed to the subject or their insurance carriers as customary. The 3.5mm circular stapler is an FDA approved product and it will also be billed to the subject or insurer in the customary fashion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 355 (Actual)
Dates: Start 2007-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ninh T Nguyen, MD, Principal Investigator — University of California, Irvine
Locations (6):
- United States (6):
  - University of California, Irvine Medical Center, Orange, California
  - Tampa General Hospital- University of South Florida, Tampa, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New York Presbyterian Hospital-Weill Cornell Medical Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited within bariatric surgery clinic at each institution
Period: Overall Study
Arm/Group | Smaller Stapler | Larger Stapler
Started | 180 | 175
Completed | 180 | 175
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smaller Stapler | Larger Stapler | Total
Number analyzed (Participants) | 180 | 175 | 355
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 175 | 355
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.1 (10.8) | 43.1 (10.1) | 43.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 138 | 273
  Male | 45 | 37 | 82
Region of Enrollment [Number; unit: participants]
  United States | 180 | 175 | 355

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Gastrointestinal Hemorrhage
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Smaller Stapler | Larger Stapler
Number analyzed (Participants) | 180 | 175
participants | 13 | 39

ADVERSE EVENTS:
Arm/Group | Smaller Stapler | Larger Stapler
Serious Adverse Events (participants affected / at risk) | 5/180 | 14/175
Other Adverse Events (participants affected / at risk) | 33/180 | 52/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smaller Stapler (N=180) | Larger Stapler (N=175)
acute renal failure (Gastrointestinal disorders) | 1 (5) | 0 (0)
anastomotic leak/intraadbdominal abscess (Gastrointestinal disorders) | 2 (5) | 2 (14)
myocardial infarction (Cardiac disorders) | 1 (5) | 0 (0)
GI obstruction (Gastrointestinal disorders) | 1 (5) | 4 (14)
pneumonia (Immune system disorders) | 0 (0) | 1 (14)
pulmonary embolism (General disorders) | 0 (0) | 2 (14)
GI hemorrhage (Gastrointestinal disorders) | 0 (0) | 5 (14)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smaller Stapler (N=180) | Larger Stapler (N=175)
GI hemorrhage (Gastrointestinal disorders) | 6 (33) | 6 (52)
anastomotic stricture (Gastrointestinal disorders) | 7 (33) | 28 (52)
cardiac arrhythmia (Cardiac disorders) | 0 (0) | 1 (52)
superficial wound infection (General disorders) | 16 (33) | 12 (52)
prolonged diarrhea (Gastrointestinal disorders) | 1 (33) | 0 (0)
peripheral neuropathy/parethesia (General disorders) | 1 (33) | 1 (52)
marginal ulcer (Gastrointestinal disorders) | 1 (33) | 3 (52)
dehydration (General disorders) | 1 (33) | 2 (52)

LIMITATIONS AND CAVEATS:
* Difficulty discerning GI bleeding attributed to the gastrojejunostomy vs gastric pouch staple-line
* Technological differences between 3.5mm vs 4.8 mm stapler
* Operative techniques varying between study sites
* Study size may be underpowered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No